CLINICAL TRIAL: NCT02606786
Title: Effectiveness of Lumbopelvic Stabilization Exercises for Pregnancy-related Low Back Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with participant recruitment and retainment
Sponsor: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Kelli Brizzolara, Assistant Professor, Texas Woman's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17919
Record Dates: First submitted 2015-03-18; First posted 2015-11-17 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Pregnancy-related Low Back Pain
Keywords: stabilization exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- stabilization exercises (Experimental): Lumbopelvic stabilization exercises have been shown to decrease pain and disability in those with low back pain. The objective of this exercise program is to recruit and train the primary stabilizing muscles of the spine in order for them to more appropriately support the spine.
  Interventions: Other: Lumbopelvic stabilization exercises

INTERVENTIONS:
Other: Lumbopelvic stabilization exercises — The objective of this exercise program is to recruit and train the primary stabilizing muscles of the spine in order for them to more appropriately support the spine.

SUMMARY:
The purpose of this study is to examine the effectiveness of lumbopelvic stabilization exercises on women who have undergone Caesarian sections on: 1) disability using the Modified Oswestry Low Back Disability Index (OSW), 2) pain according to the Numeric Pain Rating Scale (NPRS), 3) percent change of muscle thickness of the deep abdominals using ultrasound imaging, and 4) perceived improvement using the Global Rating of Change (GROC).

DETAILED DESCRIPTION:
Pregnancy-related low back pain is a very complex problem. Decreased strength and endurance in the trunk and hip muscles have been shown in those with pregnancy-related low back pain. Lumbopelvic stabilization exercises have been shown to decrease pain and disability in those with low back pain. However, there have been very few studies with post-partum women, specifically those who have undergone Caesarian section births.

The purpose of this study is to examine the effectiveness of lumbopelvic stabilization exercises on women who have undergone Caesarian sections on: 1) disability using the Modified Oswestry Low Back Disability Index (OSW), 2) pain according to the Numeric Pain Rating Scale (NPRS), 3) percent change of muscle thickness of the deep abdominals using ultrasound imaging, and 4) perceived improvement using the Global Rating of Change (GROC).

ELIGIBILITY:
Inclusion Criteria:

* Unilateral low back pain near the sacro-iliac joint (SIJ) (distal and/or lateral to L5-S1 in the buttocks) and/or symphysis pubis
* Pain onset during pregnancy or within 3 weeks of delivery
* Most recent delivery within 6-24 weeks
* At least 2/6 positive SIJ provocation tests (thigh thrust, sacral compression, sacral distraction, sacral thrust, Gaenslen's test)
* Positive active straight leg raise (ASLR) test.

Exclusion Criteria:

* Neurological signs
* Systemic disease
* Currently pregnant

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Modified Oswestry Low Back Pain Questionnaire | 4 weeks, 12 weeks
  Low back pain (LBP)-related disability

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | 4 weeks, 12 weeks
  Pain intensity
Ultrasonographic measurements | 4 weeks, 12 weeks
  Thickness of abdominal muscles at rest and with contraction
Participant perceived level of improvement | 4 weeks, 12 weeks
  Subjective rating of change in response to treatment using the Global Rating of Change Scale (GROC)

CONTACTS AND LOCATIONS:
Overall Officials: Kelli J Brizzolara, PhD, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Dallas, Texas, United States